CLINICAL TRIAL: NCT02816541
Title: Effects of Pilates-based Therapeutic Exercises on the Postural Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 886.672
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Motor Disorders
MeSH Terms: conditions — Motor Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Pelvis Retroverted (Experimental): Pilates-based therapeutic exercises performed with a posterior pelvic tilt
  Interventions: Other: Pelvis Retroverted
- Pelvis in Neutral Position (Experimental): Pilates-based therapeutic exercises performed with a neutral position of the pelvis
  Interventions: Other: Pelvis in Neutral Position
- Control Group (Active Comparator): Aerobic exercise performed on a treadmill
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Pelvis Retroverted — Pilates-based therapeutic exercises with the pelvis retroverted - Exercises executed with the retroverted pelvis, including the Footwork (toes, arched, heels, tendon stretch), Hundred, Coordination, Frog, Leg Circles (performed at the Universal Reformer apparatus ); Double Leg Stretch (performed at the Mat apparatus); Arm Spring Series (Performed at the Cadillac apparatus); The Wall Series (Performed at the Wall).
  Arms: Pelvis Retroverted
Other: Pelvis in Neutral Position — Pilates-based therapeutic exercises with the pelvis in neutral position - Exercises executed with the retroverted pelvis, including the Footwork (toes, arched, heels, tendon stretch), Hundred, Coordination, Frog, Leg Circles (performed at the Universal Reformer apparatus ); Double Leg Stretch (performed at the Mat apparatus); Arm Spring Series (Performed at the Cadillac apparatus); The Wall Series (Performed at the Wall).
  Arms: Pelvis in Neutral Position
Other: Aerobic exercise — Aerobic exercises (walking) performed on a treadmill.
  Arms: Control Group

SUMMARY:
The Pilates Method (PM) has been widely used in the daily practice of many professionals. It is well known that anticipatory postural adjustments (APAs) have a strong relation with the improvement in performance through motor control improvement. However, no studies have investigate the PM exercises performed with pelvis in different positions on the improvement of performance, APAs and these influences on motor control. This study aims to compare the effects of practicing a single session of Pilates-based therapeutic exercises with posterior pelvic tilt and neutral position of the pelvis on the APAs of elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* no history of previous abdominal or spine surgery in the last two years
* no history of low back pain in the past 2 years (as incapacitate pain lasting at least seven days)
* no neurological disorder diagnosis

Exclusion Criteria:

* significant postural asymmetry (misalignment that exceed 2 cm of the anterior superior iliac spine)

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Balance via Center of Pressure (COP) displacement assessed by force platform | change pre to post-treatment (at least 40 min)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil